CLINICAL TRIAL: NCT06025955
Title: Evaluation of Outcomes of Minimally Invasive Non- Surgical Versus Surgical Therapy in Patients With Furcation Involvement in Mandibular Molars - A Non-inferiority Randomized Controlled Trial
Brief Title: Evaluation of Outcomes of Minimally Invasive Non- Surgical Versus Surgical Therapy in Furcation Involvement.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nehaperio123
Record Dates: First submitted 2023-08-07; First posted 2023-09-06 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Furcation Defects; Open Flap Debridement; Periodontal Diseases
MeSH Terms: conditions — Furcation Defects; Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- minimally invasive non surgical therapy (Experimental): Experimental sites designated to receive non-surgical treatment will be submitted to careful subgingival debridement using curettes and ultrasonic device using 3.5 x magnification.
  Interventions: Procedure: minimally invasive non- surgical therapy
- open flap debridement (Active Comparator): Surgical technique will be used and the full-thickness flap will be minimally elevated. The granulation soft tissue will be dissected with a blade and carefully removed with curettes.
  Interventions: Procedure: open flap debridement

INTERVENTIONS:
Procedure: minimally invasive non- surgical therapy — hand and ultrasonic instrumentation will be done
  Arms: minimally invasive non surgical therapy
Procedure: open flap debridement — flap surgery will be done
  Arms: open flap debridement

SUMMARY:
The reduced rate of success experienced in the treatment of Furcation involvement (FI) seems to result from the incomplete removal of subgingival plaque and calculus in the interradicular area owing to the peculiar anatomy of the furcation space.

Regarding the therapeutic approach, although FI treated with a conservative approach may not yield the same satisfactory results as single rooted teeth; it has been shown that teeth with FI have a remarkable survival rate following conservative treatment in patients demonstrating a satisfactory plaque control. Minimally invasive techniques aim to retain the preoperative gingival architecture, create a minimal wound and gently handle soft and hard tissues. It becomes imperative to see the differences in clinical, and patient centered outcomes of minimally invasive non- surgical versus surgical technique in the management of furcation involvement in mandibulae molar.

DETAILED DESCRIPTION:
Patients will be recruited from outpatient clinic of Department of Periodontics, PGIDS, Rohtak after screening based on given inclusion and exclusion criteria. after initial session of scaling and root planing patient will be re -elevated at the and of 6 to 8 weeks those having grade 2 furcation involvement in any mandibular molar and meeting other eligibility criteria will be randomly allocated to test group and control group Test group -Experimental sites designated to receive non-surgical treatment will be submitted to careful subgingival debridement using curettes and ultrasonic device using 3.5 x magnification.

control group-Surgical technique will be followed with minimally flap reflection and incisions will be performed with papilla preservation techniques. vertical- releasing incisions will not be made, and the full-thickness flap will be minimally elevated. The granulation soft tissue will be dissected with a blade and carefully removed with curettes. The visible calculus will be carefully removed with curettes and an ultrasonic device. The flaps will be re-positioned and sutured and patient follow up 3 to 6 months .

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients with diagnosis of generalized stage 3 periodontitis (Grade A or B) with at least one mandibular molar with FI (Degree 1 or 2-according to Hamp, 1975 and Subclass A or B- according to Tarnow and Fletcher, 1984), interproximal bone coronal to the furcation fornix and root trunk length ≤ cervical two thirds of the root length as measured on a periapical radiograph.
* Full mouth plaque score < 30% after initial therapy
* Full mouth bleeding score < 30% after initial therapy
* Having undergone a course of subgingival instrumentation in the past three months

Exclusion Criteria:

* Pregnant or lactating females
* Requiring antibiotic premedication
* Received antibiotic treatment in the previous 3 months
* Previous periodontal surgery in the last 1 year
* Smokers
* Pulpal or periapical pathology
* Third molar
* Non restorable tooth
* Trauma from occlusion

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
change in horizontal clinical attachment level (HCAL) | 3 months
  change in horizontal clinical attachment level (HCAL) of the furcation as assessed
change in horizontal clinical attachment level (HCAL) | 6 months
  change in horizontal clinical attachment level (HCAL) of the furcation as assessed

SECONDARY OUTCOMES:
changes in vertical probing depth of the furcation | 3 months
  vertical probing depth will be assessed using UNC 15probe
changes in vertical probing depth of the furcation | 6 months
  vertical probing depth will be assessed using UNC 15probe
change in changes vertical clinical attachment level of furcation | 3 months
  change clinical vertical attachment will be assessed using UNC 15 probe
change in vertical clinical attachment level of furcation | 6 months
  change in vertical clinical attachment level of furcation will be assessed using UNC 15 probe
probing pocket depth (PPD)reduction | 3 months
  probing pocket depth (PPD)reduction will be calculated around the molar at 6 sites
probing pocket depth (PPD)reduction | 6 months
  probing pocket depth (PPD)reduction will be calculated around the molar at 6 sites

CONTACTS AND LOCATIONS:
Overall Officials: Neha AGGARWAL, BDS, Principal Investigator — PT BD SHARMA UHSR HARAYANA
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No